CLINICAL TRIAL: NCT02700841
Title: A Phase II Study of Enhancing Anti-Tetanus Vaccine Response After Autologous Stem Cell Transplantation
Brief Title: Enhancing Anti--Tetanus Vaccine Response After Autologous Stem Cell Transplantation
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated prematurely due to poor recruitment.
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0669-19-FB; NCI-2015-00743 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-03-02; First posted 2016-03-07 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Melphalan; Peripheral Blood Stem Cell Transplantation; Tetanus Toxoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (vaccine, CD34 transplant, DLI) (Experimental): ARM I: Patients receive 3 doses of tetanus before transplant and on days 15, and 60 post transplant.
  Interventions: Drug: Melphalan; Procedure: Peripheral Blood Stem Cell Transplantation--CD34 HSCT; Procedure: Peripheral Blood Stem Cell Transplantation--AHSCT; Biological: T Cell-Depleted Hematopoietic Stem Cell Transplantation; Biological: Tetanus Toxoid Vaccine
- Arm II (vaccine, stem cell transplant) (Active Comparator): Patients receive 3 doses of tetanus as in Arm I. Patients receive high-dose melphalan IV on day -2 and undergo AHSCT on day 0.
  Interventions: Drug: Melphalan; Procedure: Peripheral Blood Stem Cell Transplantation--AHSCT; Biological: Tetanus Toxoid Vaccine

INTERVENTIONS:
Drug: Melphalan — Given IV
  Other Names: Alkeran; L-PAM; L-Phenylalanine Mustard; Phenylalanine Mustard; Sarcolysin
Procedure: Peripheral Blood Stem Cell Transplantation--CD34 HSCT — Undergo autologous CD34 HSCT
  Other Names: PBPC Transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
  Arms: Arm I (vaccine, CD34 transplant, DLI)
Procedure: Peripheral Blood Stem Cell Transplantation--AHSCT — Undergo AHSCT
  Other Names: PBPC transplantation; Peripheral Blood Progenitor Cell Transplantation; Peripheral Stem Cell Support; Peripheral Stem Cell Transplantation
Biological: T Cell-Depleted Hematopoietic Stem Cell Transplantation — Undergo autologous CD34 HSCT
  Arms: Arm I (vaccine, CD34 transplant, DLI)
Biological: Tetanus Toxoid Vaccine — Given IM
  Other Names: Tetanus Toxoid; TT

SUMMARY:
This pilot randomized Phase II trial (10 subjects per arm) will compare immune reconstitution following transplantation of an autologous mobilized graft product to reconstitution following transplantation of a mobilized graft product followed by an autologous lymphocyte infusion collected prior to G-CSF mobilization. All subjects will receive tetanus vaccines pre and post-transplant. The primary end point will be tetanus vaccine immune responses post-transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

1. To compare the cellular and humoral vaccine response post-transplant between the two arms by performing Elisa, and T-cell enzyme-linked immunospot (ELISPOT) assays
2. To determine the feasibility and safety of this approach

SECONDARY OBJECTIVES:

1. To compare post-transplant recovery of innate and adaptive immune cells (CD8, CD4, CD19, NK, γδ T-cells), in addition to T-cell phenotype markers between the two arms.
2. To compare post-transplant recovery of T-regs and MDSCs between the two arms.
3. To compare progression free survival (PFS) at 2 years post-transplant

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 19 years to 70 years old at time of study entry (consent)
2. Diagnosis of Multiple Myeloma as per updated International Myeloma Working Group (IMWG) criteria .
3. Must have measurable disease defined as: for secretory MM, serum monoclonal protein ≥1.0 g/dL, urine monoclonal protein ≥200 mg/24 hrs, and involved free light chain ≥ 10 mg/dL; or in case of non-secretory MM, bone marrow plasma cell percentage ≥30%.
4. Must have standard risk myeloma (see exclusion criterion 4).
5. Must have received bortezomib, lenalidomide and dexamethasone (VRd) as a form of induction therapy pre-AHSCT (use of cyclophosphamide, bortezomib and dexamethasone may be allowed for up to 2 weekly doses before initiation of VRd induction, if necessary clinically for cytoreduction)
6. Able to understand and sign a consent form.
7. Creatinine clearance equal or > 60 ml/min (calculated)
8. Ejection fraction equal or > 50% before admission for transplant as per institutional standards. Patients with coronary heart disease (recent myocardial infarctions, angina, cardiac stent, or bypass surgery in the last 6 months or arrhythmia) need to be cleared by cardiology as per institutional BMT standards.
9. Serum bilirubin, ALT, AST less than 3 X upper limit of normal
10. FVC, FEV1 or DLCO >50% predicted before admission for transplant as per institutional standards. Patients on home oxygen are not allowed on the protocol.
11. No more than 6 months of pre-transplant MM chemotherapy is allowed (from the date of the start of the induction therapy).
12. KPS ≥ 70%or ECOG 0-2.
13. Must be eligible to receive Melphalan dose of 200mg/m2
14. A female of child-bearing potential, must have two negative urine pregnancy test results within 10 to 14 days prior to starting the first dose of vaccine pre-transplant as a way of ensuring safe transplant planning.

Exclusion Criteria:

1. Participation in another clinical study with an investigational product during the last 28 days.
2. Prior stem cell transplant (either autologous or allogeneic)
3. Creatinine clearance < 60 ml/min (calculated)
4. High risk MM defined as those with the following disease, fluorescence in situ hybridization and/or cytogenetic features: del17p, del1p with 1q gain, t(4;14), t(14;16), t(14;20), >1 cytogenetic abnormality on karyotype, hypodiploid, plasma cell leukemia (primary or secondary), or subjects who failed to achieve ≥PR to induction therapy (i.e. VRd) and required salvage induction prior to AHSCT.
5. Documented central nervous system or extramedullary disease.
6. Significant organ dysfunction deemed to carry inappropriate risk for AHSCT.
7. Intention or plans for cyclophosphamide mobilization.
8. Known allergic reactions after previous tetanus diphtheria vaccination or had a condition of Guillain Barre Syndrome (GBS)
9. Known active hepatitis B, C or HIV infections on initial assessment.
10. Enrollment on any other transplant related protocols.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2020-01-09 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D'Angelo, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Vaccine, CD34 Transplant, DLI) | Arm II (Vaccine, Stem Cell Transplant)
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Vaccine, CD34 Transplant, DLI) | Arm II (Vaccine, Stem Cell Transplant) | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 2 | 4 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (4.8) | 66.8 (1.7) | 64.1 (4.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 4 | 3 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Safely Treated Participants (Feasibility and Safety)
Description: Determine safety of outcomes based on the number of safely treated participants by CTCAE version 5.0 tool
Time Frame: Through 180 days post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Vaccine, CD34 Transplant, DLI) | Arm II (Vaccine, Stem Cell Transplant)
Number analyzed (Participants) | 4 | 4
Participants | 4 | 4

ADVERSE EVENTS:
Time Frame: Adverse Event Data was collected from the start of any protocol intervention to day 180 post transplant.
Arm/Group | Arm I (Vaccine, CD34 Transplant, DLI) | Arm II (Vaccine, Stem Cell Transplant)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Vaccine, CD34 Transplant, DLI) (N=4) | Arm II (Vaccine, Stem Cell Transplant) (N=4)
white blood cell decreased (Investigations) | 4 (12) | 4 (12)
Lymphocyte Count Decreased (Investigations) | 2 (6) | 3 (8)
Neutrophil Count Decreased (Investigations) | 1 (2) | 3 (5)
Platelet Count Decreased (Investigations) | 4 (11) | 2 (5)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT02700841/Prot_SAP_000.pdf